CLINICAL TRIAL: NCT01609907
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Rosuvastatin and Valsartan in Healthy Male Volunteer
Brief Title: Pharmacokinetic Drug Interaction Between Rosuvastatin and Valsartan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH14700-101
Record Dates: First submitted 2012-01-05; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension; Hyperlipidemia
Keywords: Drug interaction; YH14700; Rosuvastatin; Valsartan; Yuhan
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental)
  Interventions: Drug: Rosuvastatin+Valsartan (Sequence 1)
- Sequence 2 (Experimental)
  Interventions: Drug: Rosuvastatin+Valsartan (Sequence 2)
- Sequence 3 (Experimental)
  Interventions: Drug: Rosuvastatin+Valsartan (Sequence 3)
- Sequence 4 (Experimental)
  Interventions: Drug: Rosuvastatin+Valsartan (Sequence 4)
- Sequence 5 (Experimental)
  Interventions: Drug: Rosuvastatin+Valsartan (Sequence 5)
- Sequence 6 (Experimental)
  Interventions: Drug: Rosuvastatin+Valsartan (Sequence 6)

INTERVENTIONS:
Drug: Rosuvastatin+Valsartan (Sequence 1) — Period 1(A) Period 2(B) Period 3(C) A: Rosuvastatin 20mg (once daily for 4 consecutive days), B: Valsartan 160mg (once daily for 4 consecutive days), C: Rosuvastatin 20mg plus Valsartan 160mg (once daily for 4 consecutive days)
  Arms: Sequence 1
Drug: Rosuvastatin+Valsartan (Sequence 2) — Period 1(C) Period 2(A) Period 3(B) A: Rosuvastatin 20mg (once daily for 4 consecutive days), B: Valsartan 160mg (once daily for 4 consecutive days), C: Rosuvastatin 20mg plus Valsartan 160mg (once daily for 4 consecutive days)
  Arms: Sequence 2
Drug: Rosuvastatin+Valsartan (Sequence 3) — Period 1(B) Period 2(C) Period 3(A) A: Rosuvastatin 20mg (once daily for 4 consecutive days), B: Valsartan 160mg (once daily for 4 consecutive days), C: Rosuvastatin 20mg plus Valsartan 160mg (once daily for 4 consecutive days)
  Arms: Sequence 3
Drug: Rosuvastatin+Valsartan (Sequence 4) — Period 1(C) Period 2(B) Period 3(A) A: Rosuvastatin 20mg (once daily for 4 consecutive days), B: Valsartan 160mg (once daily for 4 consecutive days), C: Rosuvastatin 20mg plus Valsartan 160mg (once daily for 4 consecutive days)
  Arms: Sequence 4
Drug: Rosuvastatin+Valsartan (Sequence 5) — Period 1(B) Period 2(A) Period 3(C) A: Rosuvastatin 20mg (once daily for 4 consecutive days), B: Valsartan 160mg (once daily for 4 consecutive days), C: Rosuvastatin 20mg plus Valsartan 160mg (once daily for 4 consecutive days)
  Arms: Sequence 5
Drug: Rosuvastatin+Valsartan (Sequence 6) — Period 1(A) Period 2(C) Period 3(B) A: Rosuvastatin 20mg (once daily for 4 consecutive days), B: Valsartan 160mg (once daily for 4 consecutive days), C: Rosuvastatin 20mg plus Valsartan 160mg (once daily for 4 consecutive days)
  Arms: Sequence 6

SUMMARY:
The objective of this study is to compare pharmacokinetics after single oral administration of rosuvastatin and valsartan each separately versus coadministration of rosuvastatin and valsartan in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers of aged between 20 years to 50 years
* Have a body mass index (BMI) between 19kg/m2 and 27kg/m2 inclusive
* Eligible subjects with acceptable medical history, physical examination laboratory tests, ECG during screening period
* Able to follow instruction and can participate in whole procedure of the trial
* Have signed a written informed consent voluntary, prior to the any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the drug
* Anticipate having the same adult female sexual partner, who have no possibility of being pregnant or breast-feeding and take steps to prevent conception during the study

Exclusion Criteria:

* Have history of cardiovascular disorder(congestive heart failure, complications of coronary artery stenosis stroke and etc.), respiratory disorder, renal disorder(severe renal failure and etc.), liver disorder(moderate or severe liver failure and etc.) endocrine system disorder(diabetics, impaired glucose tolerance and etc.), digestive system disorder, central nervous system disorder, mental illness or malignant tumor
* Have history of gastrointestinal disease(Crohn's disease, ulcer and etc.), gastrointestinal surgery(simple appendectomy or herniotomy excluded) that can affect the absorption of the drug
* Have suffered from a clinically significant disease within 30 days prior to the first administration
* Have a known hypersensitivity or history of clinically significant hypersensitivity to drugs including the same class drugs with rosuvastatin or valsartan, or other drug(aspirin, antibiotics and etc.)
* Have genetic myopathy, family history of myopathy, or history of myopathy to drugs
* Have systolic blood pressure higher than 150mmHg or lower than 90mmHg, or diastolic blood pressure higher than 100mmHg or lower than 60mmHg, or pulse rate more than 100times/min or less than 40times/min
* Have history of drug abuse or shown positive on drug abuse during drug screening test
* Participated in any other clinical trials within 90 days prior to the first administration
* Have used any herbal medicine, prescription drug, or generic medicine within 30 days, 14 days or 7 days prior to the first administration, respectively (provided, however, if other conditions are judged to be eligible by investigators, subjects can participate in the trial)
* Donated whole blood or blood component within 60 days or 30 days prior to the first administration, respectively, or received transfusion within 30 days prior to the first administration
* Excessive alcohol drinker(> 140g/week; 1 glass of 12° wine(125mL) = 12.0g, 1 glass of 4° beer(250mL) = 8g, 0.5 bottle of soju(180mL) = 28.8g)
* Heavy smoker(> 20 cigarettes/day)
* Excessive caffeine drinker(> 4 cups/day)
* Shown positive on serum test(HBsAg, HCV Ab, HIV Ab tests)
* Subject who is judged to be ineligible by principal investigator or sub-investigator according to various reasons including their abnormal values in clinical laboratory test
* Continuous increase of liver enzyme level(AST, ALT) of unknown cause or active liver disorder patients with liver enzyme level increasing more than 3 time of normal upper limit
* Severe renal disorder patients(with creatinine clearance (Cr) < 10mL/min when calculated with Modification of Diet in Renal Disease method)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of valsartan | 18 points up to Day 4
AUCt,ss of valsartan | 18 points up to Day 4
Cmax,ss of rosuvastatin | 18 points up to Day 4
AUCt,ss of rosuvastatin | 18 points up to Day 4
t1/2 of rosuvastatin | 18 points up to Day 4

SECONDARY OUTCOMES:
Tmax,ss of valsartan | 18 points up to Day 4
t1/2 of valsartan | 18 points up to Day 4
Cmin,ss of valsartan | 18 points up to Day 4
Tmax,ss of rosuvastatin | 18 points up to Day 4
Cmin,ss of rosuvastatin | 18 points up to Day 4
t1/2 of rosuvastatin | 18 points up to Day 4
Cmax,ss of N-desmetyl rosuvastatin | 18 points up to Day 4
AUCt,ss of N-desmetyl rosuvastatin | 18 points up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Woo-Seung Huh, MD, PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Yuhan Corporation, Seoul, South Korea